CLINICAL TRIAL: NCT02401022
Title: The Study of AZD8529 for Smoking Cessation in Female Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA/VA CSP - 1032
Record Dates: First submitted 2015-03-17; First posted 2015-03-27 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Tobacco Use Disorder
Keywords: smoking; smoking cessation; cigarette
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation | interventions — AZD8529

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD8529 low dose (Active Comparator): 1.5 mg
  Interventions: Drug: AZD8529
- AZD8529 high dose (Active Comparator): 40mg
  Interventions: Drug: AZD8529

INTERVENTIONS:
Drug: AZD8529 — comparison of different dosages of drug
  Other Names: AZD-8529

SUMMARY:
To evaluate the efficacy and safety of AZD8529 for smoking cessation in female smokers.

DETAILED DESCRIPTION:
This is a 19-week, multi-center, randomized, Phase 2 clinical study comparing the efficacy of two different doses of AZD8529 (1.5 and 40 mg) in smoking cessation. Up to 2 weeks will be allowed for the Screening Period, followed by a 1-week, single-blind run-in period. At the end of Study Week 1 (on Study Day 8), medication compliance will be one of the factors used in a predictive enrichment strategy.

ELIGIBILITY:
Inclusion Criteria:

* Be a female smoker between the ages of 18 to 75 years.
* Want to quit smoking.
* Be currently (last 30 days) smoking 10 or more cigarettes per day and report less than 3 months of consecutive smoking abstinence during the past year.
* Be able, in the opinion of the site investigator (SI), to understand and follow all protocol-specified instructions and understand and provide written informed consent.
* Be willing to provide personal information for entry into a clinical trial registry.
* Agree to use and continue using at least one acceptable contraceptive method (oral contraceptives, IUDs, contraceptive implants under the skin, contraceptive rings or patches or injections, diaphragms with spermicide, condoms with spermicide, or abstinence) or, if not of childbearing potential, must fulfill one of the following criteria at screening: post-menopausal defined as amenorrhea for at least 12 months and with follicle stimulating hormone (FSH) levels in the laboratory defined post-menopausal range and/or documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy or tubal ligation verified by the Site Investigator.
* Agree not to use any other smoking behavioral intervention (self-help or formal treatment), acupuncture, or other smoking cessation pharmacotherapy during the study.
* Agree to refrain from using dietary/herbal supplements other than vitamins and minerals for 7 days prior to receiving study drug and throughout the 13-week treatment period.
* Agree to attend all required clinic appointments (including 3 eye exams) during the course of the 19-week study.

Exclusion Criteria:

* Please contact the site for more information

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shwe Gyaw, MD, Study Chair — National Institute on Drug Abuse (NIDA)
Locations (9):
- United States (9):
  - Pharmacology Research Institute, Encino, California
  - Pacific Treatment and Research Center, La Jolla, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - University of Maryland - College Park, College Park, Maryland
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Centers for the Studies of Addiction, Philadelphia, Pennsylvania
  - Virginia Commonwelath University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD8529 Low Dose: Participants received AZD8529 1.5 mg capsule orally once daily for 13 weeks
- AZD8529 High Dose: Participants received AZD8529 40 mg capsule orally once daily for 13 weeks
Period: Overall Study
Arm/Group | AZD8529 Low Dose | AZD8529 High Dose
Started | 104 | 110
Completed | 89 | 90
Not Completed | 15 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD8529 Low Dose | AZD8529 High Dose | Total
Number analyzed (Participants) | 104 | 110 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (9.34) | 47.3 (9.63) | 47.8 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 110 | 214
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 91 | 97 | 188
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 29 | 52
  White | 75 | 76 | 151
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Abstinence
Description: The number of subjects in each treatment group who are smoking abstinence during the last 4 weeks of the treatment phase (weeks 10 through 13)
Time Frame: Weeks 10 - 13
Population: Subjects who received at least one dose of AZD8529 were included in this population.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8529 Low Dose | AZD8529 High Dose
Number analyzed (Participants) | 104 | 110
Participants | 10 | 11

ADVERSE EVENTS:
Arm/Group | AZD8529 Low Dose | AZD8529 High Dose
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/104 | 3/110
Other Adverse Events (participants affected / at risk) | 74/104 | 85/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8529 Low Dose (N=104) | AZD8529 High Dose (N=110)
Pregnancy with sponteneous abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Hidrandenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Small cell lunch cancer (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8529 Low Dose (N=104) | AZD8529 High Dose (N=110)
Headache (Nervous system disorders) | 14 (18) | 24 (36)
Diarrhoea (Gastrointestinal disorders) | 6 (9) | 11 (12)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 18 (18)
Insomnia (Psychiatric disorders) | 6 (6) | 7 (7)
Weight increased (Investigations) | 3 (3) | 3 (3)
Fatigue (General disorders) | 4 (4) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (3) | 2 (2)
Pollakiuria (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Cataract (Eye disorders) | 2 (2) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Antrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Seasonal Allergy (Immune system disorders) | 2 (2) | 1 (1)
Dental care (Surgical and medical procedures) | 0 (0) | 1 (1)
Colour blindness (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (11) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less